CLINICAL TRIAL: NCT04707235
Title: ESCORT-HU Extension: European Sickle Cell Disease Cohort - Hydroxyurea - Extension
Brief Title: ESCORT-HU Extension: European Sickle Cell Disease Cohort - Hydroxyurea - Extension Study
Status: Active, not recruiting | Type: Observational
Sponsor: Theravia (Industry)
Collaborators: International Clinical Trials Association (Other)
Responsible Party: Sponsor
Other Study IDs: ESCORT-HU Extension
Record Dates: First submitted 2020-12-22; First posted 2021-01-13 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sickle cell disease patients treated with Siklos
  Interventions: Drug: Hydroxycarbamide

INTERVENTIONS:
Drug: Hydroxycarbamide — Patients, aged ≥ 2 years old, with symptomatic SCD, treated with Siklos®.
  Other Names: Siklos; Hydroxyurea

SUMMARY:
As safety information pertaining to the long-term use of HU remains incomplete in spite of the first safety study (ESCORT-HU), an extension of the latter is proposed. ESCORT-HU Extension study aims at evaluating the long-term safety of Siklos® focusing on some questions regarding its safety when used in current practice in adults and paediatric patients treated with Siklos® and followed for up to 5 years. The study will focus on the following concerns : occurrence and incidence of malignancies, leg ulcers, male fertility impairment and serious unexpected AEs causally related to Siklos®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with symptomatic SCD,
* ≥ 2 years old,
* Treated with Siklos®,
* Having been informed of the study by the investigator and consenting to participate, or whose parents or legal guardians are consenting for their child to participate.

To allow risk evaluation, participants must belong at least to one of the subpopulations defined below:

* Participants previously enrolled in ESCORT-HU who agree to participate in ESCORT-HU Extension study,
* New participants with any of the following criteria:

  * history of HU treatment for more than 5 years or
  * prepubescent over 10 years of age for girls and 13 years of age for boys at enrolment, or
  * with history of leg ulcer, or
  * pregnant women without interruption of Siklos® 3 months before the beginning of the pregnancy or,
  * males treated with Siklos® whose partner is pregnant and without discontinuation of Siklos® 3 months before the beginning of the pregnancy.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Investigators will be recruited among physicians experienced in SCD management who are the only ones authorised to initiate Siklos® treatment hence to enrol and to follow up the participants. Investigators who are already participating in ESCORT-HU study will be asked to participate in the extension study.
  Patient selection will be based on a systematic sampling technique: during the recruitment period, patients fulfilling the inclusion criteria will be informed by their initiating physician about the ESCORT-HU Extension study and enrolled in case they agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 2093 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2025-08-21 (Estimated); Study Completion 2025-08-21 (Estimated)

PRIMARY OUTCOMES:
Occurrence and incidence of the number of malignancies, leg ulcers, male fertility impairment and serious unexpected AEs causally related to Siklos® | 5 years
Occurrence and incidence of the number of leg ulcers | 5 years
Occurrence and incidence of male fertility impairment | 5 years
Occurrence and incidence of serious unexpected AEs causally related to Siklos® | 5 years

SECONDARY OUTCOMES:
Mean age of puberty | 5 years
  Document changes in fertility status in males and females
Mean number of patients with the use of a contraception, incidence of the use of semen cryopreservation and of semen analysis performed | 5 years
  Document changes in fertility status in males and females
Incidence of the use of semen cryopreservation and of semen analysis performed | 5 years
  Document changes in fertility status in males and females
Incidence of semen analysis performed | 5 years
  Document changes in fertility status in males and females
Management of Siklos® during pregnancy and outcome of pregnancy following exposure at the time of conception or at any time during the pregnancy | 5 years
  Outcome of pregnancies Following exposure to Siklos® at the time of conception (in participant and participant's partner) or at any time during the pregnancy
Frequency and reason for temporary or permanent discontinuations of Siklos® | 5 years
  Potential barriers to the compliance to the prescription of Siklos
Number of switch and combination with alternative treatment | 5 years
Measure of quality of life with SF12 questionnaire | 5 years
  Quality of life for adults SCD patients

CONTACTS AND LOCATIONS:
Overall Officials: Mariane de Montalembert, MD, PhD, Study Chair — Hospital Necker enfants malades; Frédéric Galactéros, MD, PhD, Study Chair — Henri Mondor University Hospital
Locations (87):
- France (68):
  - Amiens - Picardie Hospital Adults, Amiens
  - Amiens Picardie Hospital Children, Amiens
  - Clinique de l'Europe Amiens, Amiens
  - Angers Hospital Adults, Angers
  - Angers Hospital Center Children, Angers
  - Robert Ballanger Hospital Adults, Aulnay-sous-Bois
  - Robert Ballanger Hospital Children, Aulnay-sous-Bois
  - Avicenne Hospital Adults, Bobigny
  - Jean Verdier Hospital Children, Bondy
  - Bordeaux Hospital Adults, Bordeaux
  - Bordeaux Hospital Children, Bordeaux
  - Ambroise Paré Hospital Children, Boulogne-Billancourt
  - Tours Regional University Hospital Center Adults, Chambray-lès-Tours
  - Estaing Hospital Children, Clermont-Ferrand
  - Louis Mourier Hospital Adults, Colombes
  - Louis Mourier Hospital Children, Colombes
  - Sud Francilien Hospital Center Adults, Corbeil-Essonnes
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Sud Oise Public Hospital Group Adults, Creil
  - Henri Mondor Hospital Adults, Créteil
  - Intercommunal Hospital Center of Créteil Adults and Children, Créteil
  - Dreux Hospital Center Children, Dreux
  - Gonesse Hospital Children, Gonesse
  - Marne-La-Vallée Hospital Center Children, Jossigny
  - Grenoble Hospital Adults, La Tronche
  - Grenoble Hospital Children, La Tronche
  - Bicêtre Hospital Adults, Le Kremlin-Bicêtre
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - Jeanne De Flandre Hospital Children, Lille
  - Hôpital Saint-Vincent de Paul, Lille
  - Hôpital Mère-Enfant - CHU de Limoges, Limoges
  - Edouard Herriot Hospital Adults, Lyon
  - Hematology and oncology institute Children, Lyon
  - Timone Hospital Adults, Marseille
  - Timone Hospital Children, Marseille
  - Meaux Hospital Center Adults, Meaux
  - Meaux Hospital Center Children, Meaux
  - St Eloi Hospital Adults, Montpellier
  - Montpellier Hospital Children, Montpellier
  - Emile Muller Hospital Adults, Mulhouse
  - Nantes Hospital Children, Nantes
  - Nantes Hospital Adults, Nantes
  - Nice Hospital Children, Nice
  - Orléans Hospital Adults, Orléans
  - Armand Trousseau Hospital Children, Paris
  - Saint-Antoine Hospital Adults, Paris
  - Georges Pompidou European Hospital Adults, Paris
  - Necker Hospital Adults, Paris
  - Necker Hospital Children, Paris
  - Robert Debré Hospital Children, Paris
  - Centre hospitalier Perpignan, Perpignan
  - Poitiers Hospital Adults, Poitiers
  - American Hospital Children, Reims
  - Reims Hospital Adults, Reims
  - Pontchaillou Hospital Adults, Rennes
  - Charles Nicolle Hospital Adults, Rouen
  - Rouen Hospital Children, Rouen
  - Yves Le Foll. Hospital Center Children, Saint-Brieuc
  - Delafontaine Hospital Center Adults, Saint-Denis
  - Delafontaine Hospital Center Children, Saint-Denis
  - Saint-Quentin Hospital Center Adults, Saint-Quentin
  - Hautepierre Hospital Children, Strasbourg
  - Children Hospital, Toulouse
  - Toulouse University Institute of cancer Adults, Toulouse
  - Clocheville Regional University Hospital Center Children, Tours
  - Nancy Hospital Children, Vandœuvre-lès-Nancy
  - Versailles Hospital Center Children, Versailles
- French Guiana (4):
  - CH de Cayenne, Cayenne
  - Centre hospitalier de Kourou Children, Kourou
  - Centre Hospitalier de l'Ouest Guyanais Franck Joly Adults, Saint-Laurent-du-Maroni
  - Centre Hospitalier de l'Ouest Guyanais Franck Joly Children, Saint-Laurent-du-Maroni
- Germany (5):
  - Charité Hospital Children, Berlin
  - Düsseldorf Hospital Children, Düsseldorf
  - Freiburg Hospital Children, Freiburg im Breisgau
  - Hamburg Hospital Children, Hamburg
  - Koblenz Hospital Children, Koblenz
- Laiko General Hospital Adults, Athens, Greece
- Guadeloupe (2):
  - Hôpital RICOU - CHU Pointe-à-Pitre Abymes Children, Pointe-à-Pitre
  - Hôpital RICOU - CHU Pointe-à-Pitre Abymes, Pointe-à-Pitre
- Italy (4):
  - AUO Policlinico di Modena, Modena
  - Napoli Hospital Children, Napoli
  - Padova Hospital Children, Padua
  - Verona Hospital Children, Verona
- Martinique (2):
  - CHU Fort de France Children, Fort-de-France
  - CHU Martinique Adults, Le Lamentin
- CHU Sud Réunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No